CLINICAL TRIAL: NCT01395641
Title: A Phase I/II Clinical Trial for Treatment of Aromatic L-amino Acid Decarboxylase (AADC) Deficiency Using AAV2-hAADC
Acronym: AADC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTUH-AADC-010(200802042M)
Record Dates: First submitted 2011-06-12; First posted 2011-07-15 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2022-11

CONDITIONS: Aromatic L-amino Acid Decarboxylase (AADC) Deficiency
Keywords: Aromatic Amino Acid Decarboxylase; AADC; DDC; Gene Therapy; AAV2-AADC; Viral Vector; Gene Transfer; Aromatic L-Amino Acid Decarboxylase Deficiency
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene therapy (Experimental): Intracerebral infusion of AAV2-hAADC viral vector will be performed
  Interventions: Drug: gene therapy

INTERVENTIONS:
Drug: gene therapy — AAV2-hAADC viral vector will be injected into bilateral putamen by stereotactic surgery.
  Other Names: Intracerebral infusion of AAV2-hAADC viral vector

SUMMARY:
This Phase I/II trial is to prove the efficacy and safety of AAV2-hAADC to treat patients with AADC deficiency.

DETAILED DESCRIPTION:
Aromatic L-amino acid decarboxylase (AADC) is an enzyme responsible for the final step in the synthesis of neurotransmitters dopamine and serotonin. AADC deficiency is a rare genetic disorder. Taiwanese carry a high prevalence of AADC deficiency due to the founder mutation IVS6+4 A>T, and patients usually die before the age 5-6 years due to severe motor dysfunction.

Gene therapy with adeno-associated virus (AAV) serotype 2 (AAV2) driven human AADC (hAADC) has been tested in both animal models and Phase I clinical trials of Parkinson disease. We have done a compassionate treatment of 8 patients with AADC deficiency by AAV2-hAADC and demonstrated a result that among the treated patients, 4 could stand with support, 3 could sit with support, and there was no virus-associated toxicity. The longest follow up has exceeded 4 years.

This study is to prove the safety and efficacy of AAV2-hAADC treatment for patients with Aromatic L-amino acid decarboxylase (AADC) deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. With a confirmed diagnosis of AADC, including cerebrospinal fluid analysis to show reduced levels of neurotransmitter metabolites, HVA and 5-HIAA, and higher L-Dopa, together with more than one mutation within AADC gene.
2. Classical clinical characteristics of AADC deficiency, such as oculogyric crises, hypotonia and developmental retardation.
3. The sick child has to be over 2 years old or a head circumference big enough for surgery.
4. Participating patients must cooperate completely for all evaluations and examinations before, during and after the whole trial.
5. Parents or guardians must sign to agree on this informed consent.

Exclusion criteria

1. Significant brain structure abnormality
2. Patients with any health or neurological doubts that may increase the risk of surgery cannot join this trial. PI has the right to evaluate the feasibility of subjects for this trial based on his/her health condition.
3. Since high-level neutralizing antibodies may disturb the therapeutic effect of gene therapy, patients with anti-AAV2 neutralizing antibody titer over 1,200 folds or an ELISA OD over 1 cannot be enrolled into this trial.
4. Subjects enrolled in this clinical trial cannot take any medications that may affect this trial.

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of therapeutic effect | 12 months
  1. At one year post-surgery, neurotransmitter metabolites (HVA or HIAA) is detectable in CSF (higher than that at pre-surgery)
  2. At one year post-surgery, PDMS-II score is higher than that at pre-surgery, with an improvement over 10 points

SECONDARY OUTCOMES:
Evaluation of safety and other therapeutic effects Evaluation for the treatment safety | 12 months
  1. The absence of intracranial bleeding, which requires surgical management, after the surgery
  2. Craniotomy-induced CSF exudation
  3. The severity of post-surgery hyperactivity (if feeding is affected and then nasogastric tube is needed)
  4. Incidence of other severe adverse events (information of adverse events of all kinds and severities will be collected, including treatment-emergent adverse events).
Evaluation of secondary therapeutic effects | 5 years
  1. Weight gain
  2. Increased signal intensity of dopamine in putamen during PET imaging
  3. Increased score in other development evaluations
Exploratory endpoint | 5 years
  1. The correlation between anti-AAV2 titer and therapeutic effect
  2. The correlation between subject's age and therapeutic effect

CONTACTS AND LOCATIONS:
Overall Officials: Wuh-Liang Hwu, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tai CH, Lee NC, Chien YH, Byrne BJ, Muramatsu SI, Tseng SH, Hwu WL. Long-term efficacy and safety of eladocagene exuparvovec in patients with AADC deficiency. Mol Ther. 2022 Feb 2;30(2):509-518. doi: 10.1016/j.ymthe.2021.11.005. Epub 2021 Nov 8. PMID 34763085
- [Derived] Chien YH, Lee NC, Tseng SH, Tai CH, Muramatsu SI, Byrne BJ, Hwu WL. Efficacy and safety of AAV2 gene therapy in children with aromatic L-amino acid decarboxylase deficiency: an open-label, phase 1/2 trial. Lancet Child Adolesc Health. 2017 Dec;1(4):265-273. doi: 10.1016/S2352-4642(17)30125-6. Epub 2017 Oct 23. PMID 30169182